CLINICAL TRIAL: NCT03264144
Title: Changing Social Norms Around Smoking: A Cluster Randomized Controlled Trial to Address Tobacco Use Among Adolescents in Hong Kong
Brief Title: Address Tobacco Use Among Adolescents in Hong Kong
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Daniel Sai-Yin Ho, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17629016
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Tobacco Use
Keywords: Social norms; Adolescent; Smoking; Randomised controlled trial
MeSH Terms: conditions — Tobacco Use; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Students in the schools assigned to the intervention group will receive the intervention after the baseline survey. The intervention will be a social norms campaign involving posters, table tents, flyers and an online banner.
  Interventions: Behavioral: Social norms campaign
- Control (No Intervention): Students in the schools assigned to the control group will not receive anything during the randomised controlled trial. They will receive the intervention materials after the trial.

INTERVENTIONS:
Behavioral: Social norms campaign — Intervention messages will mainly highlight the prevalence of Hong Kong adolescents who do not smoke cigarettes and have no intention to smoke cigarettes. The messages will be conveyed to students through posters, table tents, flyers and an online banner. Posters will be posted at prominent places in schools, table tents will be placed in school canteens, flyers will be distributed to students, and the online banner will be placed at the school website. The intervention will last for 2 months.
  Arms: Intervention

SUMMARY:
This study will examine the effectiveness of a social norms campaign in correcting smoking misperceptions, reducing smoking susceptibility and changing smoking-related behaviours in Hong Kong adolescents.

DETAILED DESCRIPTION:
The study involves a behavioural intervention with social norms approaches to correct smoking misperceptions, reduce smoking susceptibility and change smoking-related behaviours in Hong Kong adolescents. A 2-arm stratified clustered randomised controlled trial (RCT) will be conducted to evaluate the effectiveness of the intervention. A total of 18 secondary schools will be randomly selected from the 5 regions in Hong Kong and invited to the RCT. The schools will then be randomly allocated to intervention or control group in the ratio of 1:1. Secondary 1 to 5 (US Grade 7 to 11) students will be invited. Students in both intervention and control group will complete a baseline survey, and the intervention group will receive the intervention after the baseline. Intervention materials includes posters and table tents at school, flyers to students, and online banner on school website. The intervention adopts social norms approaches, and will highlight the prevalence of adolescents who do not smoke and have no intention to smoke. It will last for 2 months. Both intervention and control groups will complete follow-up surveys at 3 and 9 months. The control group will receive the intervention materials after the RCT.

ELIGIBILITY:
Inclusion Criteria:

* Local secondary schools that cover grades 1-6

Exclusion Criteria:

* International secondary schools
* Special schools for adolescents with visual, hearing or other physical impairments or disabilities

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12868 (Estimated)
Dates: Start 2017-10-13 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Perceived adolescent smoking prevalence | At the time of survey
  Perceived prevalence of current smoking secondary school students in Hong Kong
Smoking susceptibility | At the time of survey
  Intention to smoke in the next 12 months, if good friends are smoking in front, and if a good friend offered a cigarette

SECONDARY OUTCOMES:
Smoking intensity | Past 30 days
  Number of smoking days in the past 30 days, average daily cigarette consumption
Intention to quit | At the time of survey
  Intention to quit
Quit attempts | Past 3 months
  Number of quit attempts

CONTACTS AND LOCATIONS:
Overall Officials: Sai Yin Ho, Dr, Principal Investigator — The University of Hong Kong
Locations (1):
- Local secondary schools, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No